CLINICAL TRIAL: NCT03111134
Title: A New Abdomen Closure Technology Based on Component Separation: a Prospective Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Xiaonan Liu, associate professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CST001
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Fascial Closure
Keywords: abdominal wound closure techniques; layered closure; component separation technique

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Abdominal Closure (No Intervention)
- New Abdominal Closure (Experimental): modified component separation technique is used to abdomen closing.
  Interventions: Procedure: modified component separation technique

INTERVENTIONS:
Procedure: modified component separation technique — a new abdomen closure technique based on component separation technique
  Arms: New Abdominal Closure

SUMMARY:
At present, open-type abdominal surgery is routine access into the abdomen. Median incision is the common choice with open-type abdominal surgery. Layered abdomen-closing is often used at the end-time of the surgery. There are some common postoperative complications, such as incision pain, surgical site infection, surgical incision dehiscence and incisional hernia. The key to reduce the incidence of postoperative complications depends on safe and reliable technology of abdomen-closing.

It's usually difficult to close the abdomen after the incisional hernia surgery, and the recurrence of incisional hernia is high. But the recurrence fell off observably when component separation technology was applied to abdomen-closing of incisional hernia.

Based on this, we hypothesis that modified-CST applied to abdomen-closing in routine abdominal surgery may improve the quality of wound-healing.

In this prospective single-blind randomized controlled trial, traditional abdomen-closing technology and modified-CST will be used to gastric cancer surgery, and the quality of wound-healing will be evaluated to confirm which kind of abdomen-closing technology better.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >18 years of age
* undergoing gastric cancer surgery
* undergoing abdominal surgery first time
* median upper abdominal incision applied (length of incision > 5cm)
* randomly select abdominal closure technique agreed by patients and family members

Exclusion Criteria:

* women who pregnant
* coagulation disorders
* undergoing immunological therapy
* undergoing chemothearphy within 2 weeks before the surgery
* undergoing Abdominal radiotherapy within 8 weeks before the surgery
* spirit disease patients
* the expecting life span less than 48 hours
* no guarantees to follow-up for 3 years
* patients with poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Class A healing rate of the surgical incision | 1 month
  Class A healing rate of the surgical incision after operation

SECONDARY OUTCOMES:
the incidence rate of incisional complications | 1 month
  the incidence rate of any incisional complications after the surgery
the time of suture to clear | 1 month
  the time of suture to clear after the surgery
hospitalization time after operation | 1 year
  hospitalization time after operation
the incidence rate of unplanned second operation | 1 month
  the incidence rate of unplanned second operation after the surgery
the incidence rate of unplanned readmission | 1 month
  the incidence rate of unplanned readmission after the surgery
the incidence rate of acute pain | 1 month
  the incidence rate of acute pain after the surgery
the mortality | 1 month
  the mortality after the surgery with any reason
the incidence rate of incisional hernia | 3 years
  the incidence rate of incisional hernia after the surgery
hospitalization costs | 3 years
  hospitalization costs for the surgery and its complications

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Liu, Ph.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China